CLINICAL TRIAL: NCT04012242
Title: Innovative Liver Elasticity, Attenuation, and Dispersion Ultrasound Study for Patients With Nonalcoholic Steatohepatitis
Brief Title: Innovative Liver Elasticity, Attenuation, and Dispersion Ultrasound Study
Acronym: iLEAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Katsutoshi Sugimoto, Associate Professor, Tokyo Medical University
Other Study IDs: TokyoMU
Record Dates: First submitted 2019-06-27; First posted 2019-07-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Nonalcoholic Steatohepatitis; Ultrasound; Elastography
Keywords: Nonalcoholic Steatohepatitis; Ultrasound; Elastography; Dispersion
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NAFLD patients who are scheduled for liver biopsy
  Interventions: Diagnostic Test: Ultrasound application

INTERVENTIONS:
Diagnostic Test: Ultrasound application — Shear wave elastography, shear wave dispersion, attenuation imaging, and intensity analysis

SUMMARY:
The objective of this study is: (1) to investigate the correlation of ultrasound parameters (SW speed, Dispersion slope, Attenuation value, Normalized Local Variance, Liver / Kidney Intensity Ratio) with the pathological parameters (fibrosis, intralobular inflammation, ballooning degeneration and steatosis); (2) to evaluate the diagnostic performance of SW speed for liver fibrosis, Dispersion slope for intralobular inflammation and Attenuation value for steatosis by comparison with the tissue diagnosis by liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Nonalcoholic fatty liver disease (NAFLD) patients who are scheduled for liver biopsy for the differential diagnosis of NASH and/or NAFLD patients who are scheduled for the MR elastography (MRE) and MRI-proton density fat friction (MRI-PDFF).
* Without a history of alcohol use, which lead to alcoholic hepatic involvement (pure alcohol below 30 g/day for male, 20 g/day for female).

Exclusion Criteria:

* Patients with endocrine disorder (hypopituitarism, growth hormone deficiency, hyperthyroidism etc.), serious nutrition disorder, and drug-induced hepatic involvement (steroid, tamoxifen, valproic acid, amiodarone etc.), which may lead to the steatosis
* Hepatitis B, Hepatitis C and HIV patients
* Primary biliary cholangitis, Primary sclerosing cholangitis, and Autoimmune hepatitis patients
* Wilson's disease, α1-antitrypsin deficiency, and hemochromatosis patients
* Malignant liver tumor, common bile duct stone, and jaundice patients
* Patients after jejunoileal bypass surgery or massive intestinal resection surgery
* Patients whose treatment changes during the period between imaging examination and liver biopsy, including medications such as antidiabetic drugs and other treatments which may change the fat deposition or inflammation of liver.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonalcoholic fatty liver disease (NAFLD) patients who are scheduled for liver biopsy for the differential diagnosis of NASH and/or NAFLD patients who are scheduled for the MR elastography (MRE) and MRI-proton density fat friction (MRI-PDFF).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of Dispersion slope for intralobular inflammation (A01 vs. A23) | At the time of examination

SECONDARY OUTCOMES:
Correlation between ultrasound parameters and the pathological parameters | At the time of examination
Diagnostic performance of SW speed for fibrosis (F0 vs. F1234, F01 vs. F234, F012 vs. F34, and F0123 vs. F4). | At the time of examination
Diagnostic performance of Normalized Local Variance for fibrosis (F0 vs. F1234, F01 vs. F234, F012 vs. F34, and F0123 vs. F4) | At the time of examination
Diagnostic performance of Normalized Local Variance for steatosis (S0 vs. S123, S01 vs. S23, and S012 vs. S3) | At the time of examination
Diagnostic performance of Dispersion slope for intralobular inflammation (A0 vs. A123, and A012 vs. A3) | At the time of examination
Diagnostic performance of Attenuation value for steatosis (S0 vs. S123, S01 vs. S23, and S012 vs. S3) | At the time of examination
Diagnostic performance of Liver/Kidney Intensity Ratio for steatosis (S0 vs. S123, S01 vs. S23, and S012 vs. S3) | At the time of examination
Diagnostic performance of the computer aided algorithm for NASH | At the time of examination
Diagnostic performance of MRI-PDFF for steatosis (S0 vs. S123, S01 vs. S23, and S012 vs. S3). | At the time of examination
Diagnostic performance of CAP for steatosis (S0 vs. S123, S01 vs. S23, and S012 vs. S3). | At the time of examination
Diagnostic performance of MRE for fibrosis (F0 vs. F1234, F01 vs. F234, F012 vs. F34, and F0123 vs. F4). | At the time of examination

CONTACTS AND LOCATIONS:
Overall Officials: Katsutoshi Sugimoto, MD, PhD, Principal Investigator — Tokyo Medical University
Locations (18):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Rocky Vista University, Parker, Colorado
  - Northwestern University, Evanston, Illinois
  - The Surgical Hospital at Southwoods, Boardman, Ohio
  - University of Washington, Seattle, Washington
- China (3):
  - SunYatSen University First Hospital, Guangzhou
  - SunYatSen University Third Hospital, Guangzhou
  - Zhejiang University No. 2 Hospital, Hangzhou
- University Paris Nord, Paris, France
- Germany (2):
  - University of Erlangen, Erlangen
  - University of Leipzig, Leipzig
- Italy (2):
  - University of Pavia, Pavia
  - Policlinico Umberto I, Univ. La Sapienza, Rome
- Japan (2):
  - Hyogo Medical University, Hyōgo
  - Kurume University, Kurume
- South Korea (2):
  - Chung-Ang University Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Charing Cross Hospital / Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Sugimoto K, Moriyasu F, Dioguardi Burgio M, Vilgrain V, Jesper D, Strobel D, Blank V, Karlas T, Grant EG, Kelahan LC, Gabriel H, Choi BI, Nishimura T, Iijima H, Dubinsky TJ, Gao J, Lee DH, Lee JY, Zhao Y, Huang P, Zeng J, Lim A, Xie X, Barr RG, Cantisani V, Ferraioli G, Sakamaki K, Itoi T, Kage M, Yano H. US Markers and Necroinflammation, Steatosis, and Fibrosis in Metabolic Dysfunction-associated Steatotic Liver Disease: The iLEAD Study. Radiology. 2024 Aug;312(2):e233377. doi: 10.1148/radiol.233377. PMID 39162633